CLINICAL TRIAL: NCT00084721
Title: A Phase I Study of Irinotecan in Combination With Fixed Dose Celecoxib in Patients With Advanced Colorectal Cancer
Brief Title: Irinotecan and Celecoxib in Treating Patients With Unresectable or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: RP 02-24; RPCI-RP-0224
Record Dates: First submitted 2004-06-10; First posted 2004-06-11 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2013-01

CONDITIONS: Colorectal Cancer; Diarrhea
Keywords: diarrhea; recurrent colon cancer; stage IV colon cancer; recurrent rectal cancer; stage IV rectal cancer; stage III colon cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Diarrhea; Colonic Neoplasms; Rectal Neoplasms | interventions — Celecoxib; Irinotecan

INTERVENTIONS:
Drug: celecoxib
Drug: irinotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as irinotecan, work in different ways to stop tumor cells from dividing so they stop growing or die. Celecoxib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Giving irinotecan with celecoxib may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of irinotecan when given with celecoxib in treating patients with unresectable or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of irinotecan when administered with celecoxib in patients with unresectable or metastatic colorectal cancer.

Secondary

* Determine the dose-limiting toxic effects and non-dose-limiting toxic effects of this regimen in these patients.
* Determine the incidence and intensity of diarrhea and myelotoxicity in patients treated with this regimen.
* Determine any responses in patients treated with this regimen.
* Determine potential mechanisms for irinotecan-induced diarrhea and protective effects of celecoxib on diarrhea prevention in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of irinotecan. Patients are assigned to 1 of 2 treatment groups.

* Group I: Patients receive a fixed dose of irinotecan IV over 90 minutes on days 1, 8, 15, and 22 and oral celecoxib twice daily on days 10-42. Courses repeat every 42 days in the absence of disease progression or unacceptable toxicity.
* Group II: Patients receive irinotecan as in group I at escalating doses and oral celecoxib twice daily on days 0-42. Treatment continues as in group I.

Cohorts of 3-6 patients receive escalating doses of irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 18-30 patients (9 for group I, 9-21 for group II) will be accrued for this study within 1-2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer

  * Metastatic or unresectable disease
* Failed first-line or second-line therapy OR recurred after receiving fluorouracil-based adjuvant chemotherapy
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* More than 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* WBC ≥ 3,000/mm^3

Hepatic

* AST and ALT ≤ 2.5 times upper limit of normal
* Bilirubin normal
* No Gilbert's disease

Renal

* Creatinine normal OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Gastrointestinal

* Able to receive oral medications
* No prior inflammatory bowel disease
* No active ulcer disease or gastritis
* No contraindications for sigmoidoscopy
* No active colostomy

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No prior allergic reaction to compounds of similar chemical or biological composition to irinotecan, celecoxib, sulfonamides, or other study agents
* No active or ongoing infection
* No other concurrent uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent filgrastim (G-CSF) or sargramostim (GM-CSF)

Chemotherapy

* See Disease Characteristics
* No more than 2 prior different chemotherapy regimens, including adjuvant therapy
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No prior irinotecan

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior radiotherapy and recovered
* No prior radiotherapy of more than 3,000 cGy
* No prior radiotherapy to extended marrow-generating fields
* No prior abdomino-pelvic irradiation

Surgery

* No prior abdominoperineal resection

Other

* More than 2 weeks since prior cyclo-oxygenase-2 (COX-2) inhibitors
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational agents
* No other anticancer therapy
* No other concurrent COX-2 inhibitors

  * Low-dose aspirin allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2005-03; Primary Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States